CLINICAL TRIAL: NCT04815083
Title: A Prospective Multi-center Clinical Study Evaluating the Use of PD G 506 A and the Eagle V1.2 Imaging System for the Visualization of Carcinoma During Breast Conserving Surgery
Brief Title: Fluorescence Imaging of Carcinoma During Breast Conserving Surgery
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated due to closure of Sponsor business
Sponsor: SBI ALApharma Canada, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: SBI-CIP 20-002
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Results first posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Breast Neoplasm Female; Breast Cancer
Keywords: Breast conserving surgery; Fluorescence Imaging; Intraoperative margin assessment
MeSH Terms: conditions — Breast Neoplasms | interventions — Aminolevulinic Acid

STUDY DESIGN:
Intervention Model Description: Part A of the study is open-label. All patients in Part A will receive the investigational drug and will undergo standard of care breast conserving surgery (BCS) followed by fluorescence-guided resection. Part B of the study is randomized and placebo controlled; patients will be randomized to receive placebo + standard of care BCS alone or PD G 506 A + SoC BCS followed by fluorescence-guided resection.
Who Masked: Participant, Outcomes Assessor
Masking Description: In Part B, the participant and pathologist will be blind to treatment arm allocation for the duration of the study. The surgeon will be blind to treatment arm allocation up until the time that standard of care resection is complete. The blind will be broken during the surgical procedure after the surgeon declares standard of care resection complete.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of Care Arm (Placebo Comparator): Patients in this arm will receive the placebo orally approximately 3 hrs prior to anesthesia followed by standard of care BCS. Fluorescence imaging will be performed on tissue specimens resected prior to completion of standard of care resection. Fluorescence-guided resection will not be performed in patients in this arm.
  Interventions: Drug: Placebo
- PD G 506 A + Fluorescence-Guided Resection Arm (Experimental): Patients in this arm will receive PD G 506 A orally approximately 3 hrs prior to anesthesia followed by standard of care BCS. Fluorescence imaging will be performed on tissue specimens resected prior to completion of standard of care resection. Fluorescence imaging performed after SoC BCS is complete will guide the resection of additional tissue.
  Interventions: Drug: Aminolevulinic Acid Hydrochloride; Device: Eagle V1.2 Imaging System

INTERVENTIONS:
Drug: Aminolevulinic Acid Hydrochloride — PD G 506 A for oral solution (aminolevulinic acid [ALA] hydrochloride [HCl] granules for oral solution) is administered as a single dose (20 mg/kg body weight) approximately 3 hours (min 2 hours, max 4 hours) prior to anesthesia.
  Other Names: PD G 506 A
  Arms: PD G 506 A + Fluorescence-Guided Resection Arm
Device: Eagle V1.2 Imaging System — Fluorescence imaging camera and associated accessories used to view and capture fluorescence and white light images and videos of the surgical cavity and excised tissue specimens during the surgical procedure.
  Arms: PD G 506 A + Fluorescence-Guided Resection Arm
Drug: Placebo — Oral placebo is administered as a single dose approximately 3 hours (min 2 hours, max 4 hours) prior to anesthesia.
  Arms: Standard of Care Arm

SUMMARY:
Breast conserving surgery (BCS) is performed on patients with breast cancer to resect and completely remove the cancer while conserving as much of the surrounding healthy tissue as possible. Current methods do not allow surgeons to determine the completeness of surgical resection in real-time. This often results in the need for a second surgical procedure, or in some cases more than two surgical procedures in order to have confidence that all cancer has been removed.

This Phase 3 study will evaluate the safety and efficacy of the fluorescent imaging agent PD G 506 A for the real-time visualization of cancer during standard of care breast conserving surgery. PD G 506 A is an investigational drug which is converted in the body into a fluorescent molecule that accumulates in cancer cells. Patients receiving PD G 506 A will undergo standard of care breast conserving surgery followed by fluorescence imaging and removal of any potentially cancerous tissue left behind in the surgical cavity.

DETAILED DESCRIPTION:
Re-operations due to positive margins following breast conserving surgery (BCS) increase poor cosmesis, complications, discomfort, stress, adjuvant delay, medical costs and risk of local recurrence. Reducing positive margin rates can be achieved through optimizing surgical procedures. This study evaluates a new method for surgeons to visualize carcinoma in real-time, both in the surgical cavity and on the margins of excised specimen(s) during the index BCS procedure.

The active ingredient of PD G 506A is aminolevulinic acid hydrochloride (ALA HCl). ALA HCl is a prodrug that is metabolized intracellularly to form the fluorescent molecule protoporphyrin IX (PpIX). The exogenous application of ALA HCl leads to a highly selective accumulation of PpIX in malignant tissues.

This Phase 3, 2-part, single-blind [pathologist(s)-blinded] randomized placebo-controlled trial study is designed to evaluate the efficacy and safety of PD G 506 A to aid in the visualization of carcinoma during BCS. The Eagle V1.2 Imaging System will be used in this trial to visualize PpIX fluorescence.

Part A is an open-label training phase of the study to optimize workflow and Part B of the study is randomized and single-blind and will serve as the pivotal portion of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Female, 18 years or older
2. Histologically or cytologically confirmed primary breast cancer (includes invasive lobular carcinoma, invasive ductal carcinoma, inflammatory breast cancer, papillary breast cancer, adenoid cystic carcinoma of the breast, mucinous breast cancer, metaplastic breast cancer, cribriform carcinoma and ductal carcinoma in situ, alone or in combination with invasive disease)
3. Scheduled for a lumpectomy (including bilateral lumpectomy) of a breast malignancy (eligibility for breast conserving surgery/partial mastectomy based on clinical staging using TNM staging system (AJCC Cancer Staging Manual: Breast Cancer, 8th Edition70).
4. Patient must have normal organ and bone marrow function and be appropriate surgical candidate per site standard of care
5. Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) starting the day entering the study, and for the duration of the study period (until the Week 2 visit)

Exclusion Criteria:

1. Currently on (neo)adjuvant therapy to treat another cancer
2. Receiving or intended to receive neoadjuvant therapy to treat the primary breast cancer (including chemotherapy, endocrine therapy and radiotherapy)
3. Stage 4 cancer, inclusive of metastatic disease
4. Non-invasive diseases of the breast (includes lobular carcinoma in situ, phyllodes and Paget's disease of the breast)
5. Patients who have had the following procedures performed on the involved breast:

   1. Surgery for a benign lesion(s) within 1 year of the BCS date
   2. Breast implants inserted within 1 year of the BCS date
   3. Breast reduction, surgery for malignant disease or mastectomy (at any time prior to the BCS date)
   4. Surgery for a benign lesion(s) or insertion of implants >1 year prior to the BCS date and who have signs of ongoing inflammation, active tissue healing and/or extensive scarring
   5. Radiation at any time prior to the BCS date and who have signs of ongoing inflammation, active tissue healing and/or extensive scarring
6. Patients for whom intraoperative frozen section analysis is planned
7. Patients who have not recovered from adverse events due an investigational pharmaceutical or diagnostic agents administered more than 30 days prior to their scheduled surgical procedure
8. History of hypersensitivity to ALA HCl or porphyrins
9. Known or documented personal or family history of porphyria
10. Patient has a recording of any parameter as defined below:

    1. Bilirubin: Above upper limit of normal
    2. Aspartate aminotransferase (SGOT): > 2.5 X institutional upper limit of normal
    3. Alanine aminotransferase ( (SGPT): > 2.5 X institutional upper limit of normal
11. Patient has serum creatinine >1.5 times institutional upper limit of normal, OR calculated creatinine clearance > 60 mL/min/1.73 m² for patients with creatinine levels above institutional normal.
12. Uncontrolled concurrent illness, that in the opinion of the Investigator would prevent the patient from participation in the study, including but not limited to:

    1. Ongoing or active infection;
    2. Cardiovascular disease (e.g. symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia).
13. Patients who have the following collagen vascular diseases:

    1. Lupus
    2. Scleroderma
14. Use of an investigational drug within 30 days of their scheduled surgical procedure
15. Simultaneous use of other potentially phototoxic substances (such as St. John's wort, griseofulvin, thiazide diuretics, sulfonylureas, phenothiazines, sulphonamides, quinolones and tetracyclines), and topical preparations containing ALA for 24 hours during the perioperative period.
16. Social or medical situations including uncontrolled psychiatric illnesses that would in the opinion of the Investigator limit compliance with study requirements (e.g. ability to travel for follow-up)
17. Patients who are pregnant or become pregnant (it is unknown if ALA HCl is teratogenic or has abortifacient effects)
18. Patients who are breast feeding (there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ALA HCl, breastfeeding should be discontinued if the mother is treated with ALA HCl)
19. Inability to consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2024-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph DaCosta, PhD, Study Director — SBI ALApharma Canada
Locations (7):
- United States (7):
  - Stamford Hospital, Stamford, Connecticut
  - BayCare Morton Plant Hospital, Clearwater, Florida
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Orlando Health, Inc., Orlando, Florida
  - BayCare St. Joseph's Hospital, Tampa, Florida
  - Montefiore Medical Center, The Bronx, New York
  - Aurora St. Luke's Medical Centre, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between 04/27/2021 and 08/30//2025. Patients were recruited by their surgeon at surgical clinic visits. Participants were recruited at each of the 7 study sites.
Pre-assignment Details: Fifty-seven (57) patients were enrolled for baseline characteristics as indicated in eligibility criteria prior to assignment in Part A of the study. Four (4) enrolled patients were excluded after enrollment due not meeting eligibility requirements. Three (3) patients who were enrolled were not completed due to a physician decision (1 patient) or a study pause (2 patients). The Part B (randomized and placebo controlled) was never initiated. The trial was terminated beforehand.
Period: Overall Study
Arm/Group | PD G 506 A + Fluorescence-Guided Resection Arm
Started | 57
PD G 506 A + Fluorescence-Guided Resection Arm | 50
Completed (Participants were recruited exclusively for Part A. Participants completed the study in full accordance with the protocol, before data collection for the endpoints in Part B.) | 50
Not Completed | 7
Not completed — Physician Decision | 1
Not completed — Study pause | 2
Not completed — Screening failure | 4

BASELINE CHARACTERISTICS:
Population: The aim of Part A of the study is to provide training to the participating sites on the study procedures, and to determine the final number of subjects required for analysis of the endpoints in Part B of the study. The study was terminated early after the completion of Part A and before the start of Part B.
Groups:
- PD G 506 A + Fluorescence-Guided Resection (Part A): Patients in this arm received PD G 506 A orally approximately 3 hrs prior to anesthesia followed by standard of care BCS. Fluorescence imaging was be performed on tissue specimens resected prior to completion of standard of care resection. Fluorescence image-guided resection was performed after SoC BCS was complete.
Arm/Group | PD G 506 A + Fluorescence-Guided Resection (Part A)
Number analyzed (Participants) | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 35
  >=65 years | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13
  Not Hispanic or Latino | 43
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 39
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  United States | 57
Diagnosis [Count of Participants; unit: Participants]
  Invasive carcinoma (± in situ carcinoma) | 39
  In situ carcinoma | 13
  Other (± in situ carcinoma) | 4
  Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Positive Margin Conversion Rate
Description: Percentage of patients with negative-margins following fluorescence-guided resection (FGR) among patients all patients imaged
Time Frame: 2 weeks
Population: The study was terminated early after the completion of Part A, before data collection for the analysis of the endpoints in Part B had begun, as per the protocol. The only objectives of Part A were to conduct training for the participating trial sites and to optimize the study workflow for Part B, so this endpoint will not be analysed.
Groups:
- PD G 506 A + Fluorescence-Guided Resection Arm (Part A): Patients in this arm will receive PD G 506 A orally approximately 3 hrs prior to anesthesia followed by standard of care BCS. Fluorescence imaging will be performed on tissue specimens resected prior to completion of standard of care resection. Fluorescence imaging performed after SoC BCS is complete will guide the resection of additional tissue.
  Aminolevulinic Acid Hydrochloride: PD G 506 A for oral solution (aminolevulinic acid [ALA] hydrochloride [HCl] granules for oral solution) is administered as a single dose (20 mg/kg body weight) approximately 3 hours (min 2 hours, max 4 hours) prior to anesthesia.
  Eagle V1.2 Imaging System: Fluorescence imaging camera and associated accessories used to view and capture fluorescence and white light images and videos of the surgical cavity and excised tissue specimens during the surgical procedure.
Arm/Group | PD G 506 A + Fluorescence-Guided Resection Arm (Part A)
Number analyzed (Participants) | 0

2. Primary Outcome: Diagnostic Performance (Specificity)
Description: Patient-level specificity to identify residual carcinoma
Time Frame: 2 weeks
Population: as for outcome 1
Arm/Group | PD G 506 A + Fluorescence-Guided Resection Arm (Part A)
Number analyzed (Participants) | 0

3. Primary Outcome: Diagnostic Performance (Sensitivity)
Description: Patient-level sensitivity to identify residual carcinoma
Time Frame: 2 weeks
Population: as for outcome 1
Arm/Group | PD G 506 A + Fluorescence-Guided Resection Arm (Part A)
Number analyzed (Participants) | 0

4. Secondary Outcome: Orientation-level Diagnostic Performance
Description: Orientation-level diagnostic performance of PD G 506 A-induced fluorescence to determine the presence or absence of cancer in the surgical cavity as compared to margin histopathology.
Time Frame: 2 weeks
Population: as for outcome 1
Arm/Group | PD G 506 A + Fluorescence-Guided Resection Arm (Part A)
Number analyzed (Participants) | 0

5. Secondary Outcome: Positive Margin Conversion Rate Among All Patients
Description: Percentage of patients with at least one histopathology-positive margin following SoC who then have ALL histopathology-negative margins following FGR, among all patients imaged.
Time Frame: 2 weeks
Population: as for outcome 1
Arm/Group | PD G 506 A + Fluorescence-Guided Resection Arm (Part A)
Number analyzed (Participants) | 0

6. Secondary Outcome: Patient-level Diagnostic Performance
Description: Patient-level sensitivity, specificity, NPV, PPV of PD G 506 A-induced fluorescence to determine the presence or absence of residual cancer.
Time Frame: 2 weeks
Population: as for outcome 1
Arm/Group | PD G 506 A + Fluorescence-Guided Resection Arm (Part A)
Number analyzed (Participants) | 0

7. Secondary Outcome: Patient-level Diagnostic Performance of PD G 506 A to Detect Residual Cancer at the End of FGR With Modified Patient-level Definitions
Description: Patient-level sensitivity, specificity, PPV and NPV to determine the presence or absence of residual cancer in the surgical cavity at the end of FGR (using modified patient-level definitions).
Time Frame: 2 weeks
Population: as for outcome 1
Arm/Group | PD G 506 A + Fluorescence-Guided Resection Arm (Part A)
Number analyzed (Participants) | 0

8. Secondary Outcome: Patient-level Diagnostic Performance of PD G 506 A to Detect Cancer After SoC BCS
Description: Patient-level sensitivity, specificity, PPV and NPV to determine the presence or absence of cancer in the surgical cavity after SoC BCS.
Time Frame: 2 weeks
Population: as for outcome 1
Arm/Group | PD G 506 A + Fluorescence-Guided Resection Arm (Part A)
Number analyzed (Participants) | 0

9. Secondary Outcome: Patient-level Diagnostic Performance of PD G 506 A to Detect Cancer After SoC With Modified Patient-level Definitions
Description: Patient-level sensitivity, specificity, PPV and NPV to determine the presence or absence of cancer in the surgical cavity after SoC (using modified patient-level definitions).
Time Frame: 2 weeks
Population: as for outcome 1
Arm/Group | PD G 506 A + Fluorescence-Guided Resection Arm (Part A)
Number analyzed (Participants) | 0

10. Secondary Outcome: Patient-level False Negative Rate of at the End of FGR
Description: Percentage of patients assessed as residual tumor negative at the end of FGR who had positive final margins on histopathology.
Time Frame: 2 weeks
Population: as for outcome 1
Arm/Group | PD G 506 A + Fluorescence-Guided Resection Arm (Part A)
Number analyzed (Participants) | 0

11. Secondary Outcome: Patient-level False Positive Rate
Description: Percentage of patients in whom SOC final margins were carcinoma negative and all FL-driven shave specimens are carcinoma-negative.
Time Frame: 2 weeks
Population: as for outcome 1
Arm/Group | PD G 506 A + Fluorescence-Guided Resection Arm (Part A)
Number analyzed (Participants) | 0

12. Secondary Outcome: Patients With Carcinoma-negative Margins After SoC Found to Have Residual Tumor Following SoC That Was Identified With FL Imaging
Description: Percentage of patients with histopathology-negative margins at the end of SoC who have at least one orientation that was both FL-positive and histopathology-positive among (1) patients with histopathology negative final margins after SOC and (2) all patients imaged.
Time Frame: 2 weeks
Population: as for outcome 1
Arm/Group | PD G 506 A + Fluorescence-Guided Resection Arm (Part A)
Number analyzed (Participants) | 0

13. Secondary Outcome: Patient-level True Negative Rate at the End of SoC
Description: Percentage of patients with no fluorescence identified at the end of SoC in whom all final margins after SoC are histopathologically confirmed to be negative for carcinoma.
Time Frame: 2 weeks
Population: as for outcome 1
Arm/Group | PD G 506 A + Fluorescence-Guided Resection Arm (Part A)
Number analyzed (Participants) | 0

14. Secondary Outcome: Patient-level Diagnostic Performance to Identify in Vivo Residual Carcinoma After FGR
Description: Patient-level in vivo diagnostic performance of PD G 506 A-induced fluorescence to determine the presence or absence of residual cancer in the surgical cavity at the end of FGR as compared to the final margin histopathology.
Time Frame: 2 weeks
Population: as for outcome 1
Arm/Group | PD G 506 A + Fluorescence-Guided Resection Arm (Part A)
Number analyzed (Participants) | 0

15. Secondary Outcome: Orientation Discordant Fluorescence Status
Description: Percentage of orientations where in vivo and ex vivo fluorescence assessments are discordant.
Time Frame: 2 weeks
Population: as for outcome 1
Arm/Group | PD G 506 A + Fluorescence-Guided Resection Arm (Part A)
Number analyzed (Participants) | 0

16. Secondary Outcome: Patient-level Re-operation Rate
Description: Percentage of patients receiving a 2nd surgery on the ipsilateral breast within 1 year of index BCS to remove suspected residual disease.
Time Frame: 1 year
Population: as for outcome 1
Arm/Group | PD G 506 A + Fluorescence-Guided Resection Arm (Part A)
Number analyzed (Participants) | 0

17. Secondary Outcome: Patient-level Early Re-operation Rate
Description: Percentage of patients receiving an early 2nd surgery (planned or actual) on the ipsilateral breast related to positive final margins.
Time Frame: 3 - 6 months
Population: as for outcome 1
Arm/Group | PD G 506 A + Fluorescence-Guided Resection Arm (Part A)
Number analyzed (Participants) | 0

18. Secondary Outcome: Amount of Tissue Removed With FGR Beyond SoC
Description: Weight (mg) of all tissue removed based on SoC and/of FGR.
Time Frame: 3 - 6 months
Population: as for outcome 1
Arm/Group | PD G 506 A + Fluorescence-Guided Resection Arm (Part A)
Number analyzed (Participants) | 0

19. Secondary Outcome: Patient Satisfaction With Breast
Description: Patient satisfaction with the cosmetic outcome of breast conserving surgery performed based on SoC in combination with PD G 506 A and the Eagle V1.2 Imaging System.
Time Frame: 2 weeks, 3-, 6- and 12-months
Population: as for outcome 1
Arm/Group | PD G 506 A + Fluorescence-Guided Resection Arm (Part A)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: All adverse events were followed from the time of consent to through to the Week 2 visit (~14 days after surgery). If a serious or non-serious adverse event (AE) was recorded at the Week 2 visit, the participant was assessed for an additional 7 days for non-serious adverse events or for at least an additional 30 calendar days for serious adverse events following the Week 2 visit. Any serious adverse events were followed until resolution or stabilization.
Arm/Group | PD G 506 A + Fluorescence-Guided Resection Arm (Part A)
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 1/50
Other Adverse Events (participants affected / at risk) | 16/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PD G 506 A + Fluorescence-Guided Resection Arm (Part A) (N=50)
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PD G 506 A + Fluorescence-Guided Resection Arm (Part A) (N=50)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 4 (5)
Procedural pain (Injury, poisoning and procedural complications) | 8 (10) — Post-operative pain in affected breast
Nausea (Gastrointestinal disorders) | 6 (6)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
Study was terminated early prior to meeting expected enrolment for Part A. No formal data analysis was performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-11): https://cdn.clinicaltrials.gov/large-docs/83/NCT04815083/Prot_SAP_001.pdf